CLINICAL TRIAL: NCT00796549
Title: A Phase II Single-arm Trial of BIBW 2992 in EGFR FISH Positive Non-small Cell Lung Cancer Patients
Brief Title: BIBW2992 (Afatinib) in Advanced (EGFR-FISH +) NSCLC (Non Small Cell Lung Cancer) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.40; 2008-001264-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental): BIBW 2992 in EGFR FISH positive NSCLC patients
  Interventions: Drug: BiBW 2992

INTERVENTIONS:
Drug: BiBW 2992 — BIBW 2992 in EGFR FISH positive NSCLC patients

SUMMARY:
The primary objective of this open-label, single arm Phase II trial is to explore the efficacy of BIBW 2992 defined by the objective response rate (CR, PR) as determined by the RECIST criteria in patients with EGFR FISH positive advanced NSCLC Stage IIIB or IV, selected according to the following scheme:

* Forty (40) 1st line patients
* Thirty (30) 2nd line patients Patients entered into the trial will be treated and followed until death or lost to follow-up. Additional information will be obtained on the safety profile and PK analysis of BIBW 2992.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients aged >18 years.
2. Patients with pathologically confirmed diagnosis of NSCLC Stage IIIB (with pleural effusion) or Stage IV and histopathological classification of adeno- or bronchoalveolar carcinoma (BAC).
3. Increased EGFR gene copy number assessed by FISH analysis. After signed informed consent, positive result to EGFR FISH determination is mandatory to proceed to other screening assessments.
4. At least one tumour lesion that can accurately be measured by computed tomography (CT) or magnetic resonance imaging (MRI) in at least one dimension with longest diameter to be recorded as more or same 20 mm using conventional techniques or moro or same 10 mm with spiral CT scan.
5. Patients not previously exposed to chemotherapy for NSCLC (1st line patients, 40 in total; for these subjects adjuvant chemotherapy is allowed if at least 12 months elapsed since last course of treatment), or patients with relapse after one systemic treatment (2nd line patients, 30 in total; if less than 12 months elapsed since adjuvant chemotherapy, patients are 2nd line ones, as adjuvant chemotherapy must be considered a line of treatment).
6. Life expectancy of at least three (3) months.
7. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score 0, 1 or 2.
8. Written informed consent that is consistent with ICH-GCP guidelines.

Exclusion criteria:

1. More than two (2) prior cytotoxic chemotherapy treatment regimens for relapsed or metastatic NSCLC, included adjuvant chemotherapy if relapse occurred less than 12 months before
2. Previous treatment with erlotinib (Tarceva®), gefitinib (Iressa®) or any other EGFR inhibiting small molecule or antibody.
3. Active brain metastases (stable <4 weeks, symptomatic, requiring treatment with anticonvulsants, or leptomeningeal disease). Dexamethasone therapy will be allowed if administered as a stable dose for at least one month before randomization.
4. Chemo-, hormone- (other than megestrol acetate or steroids required for maintenance non-cancer therapy) or immunotherapy within the past 4 weeks before first drug administration.
5. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn disease, malabsorption, or CTCAE Grade >2 diarrhea of any etiology at baseline
6. Patients who have any other life-threatening illness or organ system dysfunction which, in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
7. Other malignancies diagnosed within the past five (5) years (other than non melanomatous skin cancer and in situ cervical cancer).
8. Radiotherapy within the past 2 weeks prior to treatment with the trial drug.
9. Patients with any serious active infection (i.e., requiring an IV antibiotic, antifungal, or antiviral agents).
10. Patients with known HIV, active hepatitis B or active hepatitis C.
11. Known or suspected active drug or alcohol abuse.
12. Women of child-bearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial.
13. Pregnancy or breast feeding.
14. Patients unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- Italy (13):
  - 1200.40.39011 Boehringer Ingelheim Investigational Site, Arezzo
  - 1200.40.39007 Boehringer Ingelheim Investigational Site, Aviano (PN)
  - 1200.40.39013 Boehringer Ingelheim Investigational Site, Faenza (RA)
  - 1200.40.39003 Boehringer Ingelheim Investigational Site, Genova
  - 1200.40.39010 Boehringer Ingelheim Investigational Site, Livorno
  - 1200.40.39012 Boehringer Ingelheim Investigational Site, Lugo (RA)
  - 1200.40.39008 Boehringer Ingelheim Investigational Site, Modena
  - 1200.40.39005 Boehringer Ingelheim Investigational Site, Monza (MI)
  - 1200.40.39006 Boehringer Ingelheim Investigational Site, Padua
  - 1200.40.39002 Boehringer Ingelheim Investigational Site, Perugia
  - 1200.40.39004 Boehringer Ingelheim Investigational Site, Prato
  - 1200.40.39009 Boehringer Ingelheim Investigational Site, Ravenna
  - 1200.40.39001 Boehringer Ingelheim Investigational Site, Rozzano (MI)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on December 23rd 2008 . Last patient enrolled on September 1st 2011. Patients were recruited in Oncology departments of Italian investigational sites
Groups:
- Afatinib 50mg: Afatinib 50mg film coated tablets was administered once daily as long as they were tolerated by patients, until disease progression (according to the response evaluation criteria in solid tumors)
Period: Overall Study
Arm/Group | Afatinib 50mg
Started | 218 (Excluding duplicate records for 5 patients who were screened twice)
Entered | 69 (entered and treated)
Completed | 0
Not Completed | 218
Not completed — Adverse Event | 11
Not completed — not entered | 149
Not completed — Other | 2
Not completed — Progressive disease | 56

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Objective Response
Description: Percentage of participants with best objective response: confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.0.
Time Frame: Tumour assessments were performed at baseline (tumour assessment obtained within 4 weeks prior to beginning of treatment), week 8, and every 8 weeks until last response assessment 28NOV12.
Population: Treated set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
percentage of participants | 13.0 [6.1 to 23.3]

2. Secondary Outcome: Number of Participants With Objective Response (OR) Categorized by Time
Description: Cumulative number of participants with objective response by time points with responders.
Time Frame: as for outcome 1
Population: Treated set (TS).
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
percentage of participants
  by week 8 | 11.6
  by week 96 | 13.0

3. Secondary Outcome: Duration of Confirmed Objective Response (OR)
Description: Duration of confirmed Objective Response is measured from the time of first Objective Response (OR) to the time of progression or death (or date of censoring for progression free survival).
Time Frame: as for outcome 1
Population: Treated set (TS).
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Weeks | 45.5 (36.5)

4. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: Percentage of participants with Objective response (OR) or stable disease (SD) as determined by RECIST version 1.0.
Time Frame: Every 8 weeks until last response assessment 28NOV12
Population: Treated set (TS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
percentage of participants | 50.7 [38.4 to 63.0]

5. Secondary Outcome: Duration of Confirmed Disease Control
Description: Duration of Disease Control is measured from the time of first Objective Response to the time of progression or death (or date of censoring for progression free survival) or respectively for SD as the time from date of randomization to date that disease progression.
Time Frame: Every 8 weeks until last response assessment 28NOV12
Population: Treated set (TS).
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Weeks | 37.4 (35.6)

6. Secondary Outcome: Progression Free Survival (PFS) Time
Description: Progression Free Survival time defined as time from the start of treatment to the earliest of progression (RECIST), clinical progression (investigator), start of new anti-cancer treatment or death.
Time Frame: Every 8 weeks until last response assessment 28NOV12
Population: Treated set (TS).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Weeks | 8.43 [7.43 to 15.71]

7. Secondary Outcome: Overall Survival (OS) Time
Description: Overall survival time is defined as time from the date of start of treatment to the date of death.
Time Frame: Baseline until last vital status assessment 17JUN13
Population: Treated set (TS).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Weeks | 50.43 [33.43 to 64.00]

8. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady State on Day 15 (Cpre,ss,15)
Description: Cpre,ss,15 represents the pre-dose concentration of afatinib in plasma at steady state on day 15.
Time Frame: Day 15
Population: Pharmacokinetic set (PK set) contains all patients who received study medication and have evaluable pharmacokinetic parameter data.
  Data from patients who received the starting dose of 50 mg afatinib and were still on treatment and not dose-reduced on Day 15 are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 50mg 1st Line: Afatinib 50mg film coated tablets was administered once daily as long as they were tolerated by patients, until disease progression (according to the response evaluation criteria in solid tumors). Only Patients with 1st line anti cancer treatment, indicating that they had not received prior treatment with chemotherapy.
- Afatinib 50mg 2nd Line: Afatinib 50mg film coated tablets was administered once daily as long as they were tolerated by patients, until disease progression (according to the response evaluation criteria in solid tumors). Only Patients with 2nd line anti cancer treatment, indicating that they had received one prior anti cancer treatment with chemotherapy.
Arm/Group | Afatinib 50mg 1st Line | Afatinib 50mg 2nd Line
Number analyzed (Participants) | 28 | 17
ng/mL | 37.9 (64.5) | 29.7 (61.6)

9. Secondary Outcome: Number of Participants With Clinical Relevant Finding in Gastrointestinal and Skin Disorder
Description: The safety of patients was overall assessed in terms of adverse events (AEs), graded according to US NCI CTCAE version 3.0 [R04-0474], including skin reactions and gastrointestinal AEs.
Time Frame: First administration of trial medication until 28 days after last administration of trial medication, up until 194 weeks
Population: Treated Set (TS).
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
Percentage of participants
  Diarrhoea | 82.6
  Stomatitis | 13.0
  Nausea | 14.5
  Vomiting | 13.0
  Constipation | 7.2
  Abdominal pain | 5.8
  Abdominal pain upper | 2.9
  Cheilitis | 2.9
  Dyspepsia | 2.9
  Dysphagia | 2.9
  Abdominal distension | 1.4
  Dry mouth | 1.4
  Flatulence | 1.4
  Gastritis erosive | 1.4
  Odynophagia | 1.4
  Peritoneal haemorrhage | 1.4
  Rectal haemorrahage | 1.4
  Tongue Ulceration | 1.4
  Rash | 73.9
  Skin exfoliation | 15.9
  Dry skin | 14.5
  Nail disorder | 13.0
  Pruritus | 13.0
  Dermatitis acneiform | 5.8
  Alopecia | 1.4
  Granuloma skin | 1.4
  Hirsutism | 1.4
  Hypertrichosis | 1.4
  Nail discolouration | 1.4
  Night sweats | 1.4
  palmar-plantar erythrodysaesthesia syndrome | 1.4
  Skin fissures | 1.4
  Skin reaction | 1.4

10. Secondary Outcome: Number of Participants With Clinical Relevant Findings in Laboratory Safety Parameters, Vital Signs and Left Ventricular Ejection Fraction
Description: Number of participants with clinical relevant findings in Laboratory safety parameters, vital signs and Left ventricular ejection fraction . Relevant findings or worsenings of baseline conditions were reported as Adverse Events.
  There were no clinically relevant finding reported for Vital signs and Left ventricular ejection fraction (LVEF).
Time Frame: as for outcome 9
Population: Treated Set (TS).
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
percentage of participants
  Alanine aminotransferase increased | 2.9
  Aspartate aminotransferase increased | 2.9
  Blood alkaline phosphatase increased | 2.9
  Blood bilirubin increased | 1.4
  Blood Creatine phosphokinase increased | 1.4
  Blood lactate dehydrogenase increased | 1.4
  Ejection fraction decreased | 1.4
  Gamma-glutamyltransferase increased | 1.4
  International normalised ratio increased | 1.4
  Transaminases increased | 2.9
  Weight decreased | 7.2

11. Secondary Outcome: Assessment of Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Performance status assessed according to Eastern Cooperative Oncology Group (ECOG) performance status based on categories defined below :
  0 : Fully active, able to carry on all pre-disease performance without restriction.
  1. : Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. : Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. : Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. : Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. : Dead.
  Note: The ECOG scores presented are assessed at the end of treatment not at baseline, hence the patients having ECOGs>2 are included.
Time Frame: End Of Treatment, up until 190 weeks
Population: Treated set (TS).
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 69
percentage of participants
  0 | 23.2
  1 | 40.6
  2 | 7.2
  3 | 1.4
  4 | 1.4
  Missing | 26.1

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication, up until 194 weeks
Groups:
- Afatinib 50mg: Afatinib 50mg film coated tablets where administered once daily as long as they were tolerated by patients, until a disease progression (according to the response evaluation criteria in solid tumors)
Arm/Group | Afatinib 50mg
Serious Adverse Events (participants affected / at risk) | 35/69
Other Adverse Events (participants affected / at risk) | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Gastritis erosive (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 2
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Superior vena cava syndrome (Vascular disorders) | 2
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 4
Conjunctivitis (Eye disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 53
Nausea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 4
Fatigue (General disorders) | 19
Mucosal inflammation (General disorders) | 20
Pyrexia (General disorders) | 13
Cystitis (Infections and infestations) | 5
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 51
Skin exfoliation (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.